CLINICAL TRIAL: NCT03673176
Title: Lung Volume Reduction for Severe Emphysema by Stereotactic Ablative Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Principal Investigator, Joseph B. Shrager, MD, Professor and chief of thoracic surgery division, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-protocol 23203
Record Dates: First submitted 2017-11-20; First posted 2018-09-17 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Ablative Radiotherapy (Experimental): Experimental stereotactic ablative radiation treatment
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — The prescribed dose will be 45 Gy in three fractions of 15 Gy, on each side that is treated.

SUMMARY:
Since medical therapies offer only modest palliation and minimal hopes for improved survival to COPD patients, surgical therapies have been designed that may provide greater benefits in selected patients. Lung transplantation, for example, clearly improves survival and quality of life in patients with end stage COPD. This comes at substantial economic cost, however, as well as the at the cost of complications that may result from the complex surgery and from life-long immunosuppression. In addition, nearly all lung transplants will fail within 5 years as a result of progressive bronchiolitis obliterans, which we currently have no way to prevent or treat.

A second operation designed to treat severe COPD patients is lung volume reduction surgery (LVRS). This operation, designed for patients with predominant emphysema rather than chronic bronchitis, is among the most carefully studied operations ever developed.

We believe that by reducing the volume of emphysematous lung with the precise target localization made possible by image-guided SABR, that we will be able to duplicate the benefits of surgical lung volume reduction with far less risk. We believe that this may represent a major advance in the therapy of emphysema - a highly prevalent disease. It may provide not only palliation but also increased survival, as does surgical lung volume reduction, in carefully selected patients.

DETAILED DESCRIPTION:
Stereotactic Ablative Radiotherapy (SABR), also called stereotactic body radiation therapy (SBRT), is a relatively recent advance in radiotherapy which allows high doses of radiation to be transmitted to focused areas (typically malignancies), allowing higher rates of tumoricidal activity, generally lower complications, and greater convenience for patients since it can be delivered in 1 to just a few sessions. As the radiation is administered from multiple directions according to stereotactic planning, high doses can be delivered to the tissues with rapid fall-off to relatively low doses in even nearby, surrounding normal tissues. This technique was initially applied to brain tumors- an application which over the years has met with great success. More recently, it has been applied with substantial success and is gaining increasing acceptance as a primary mode of therapy for stage I lung malignancies, and malignancies in multiple other body areas.

In the lung, the rate of pneumonitis resulting from SABR is far lower than the rates incurred by conventional external beam radiotherapy. In conventional external beam radiotherapy reported pneumonitis rates range from 13-37% (7), depending on dose and field size. Reported rates of symptomatic pneumonitis after lung SABR are significantly lower and generally are ~5% (8). SABR does, however, typically leave a scar in the area of lung that has been treated (9). Importantly, there appears to be contraction of surrounding lung parenchyma into this scar resulting in an effect that is essentially a "lung volume reduction." One often sees clear loss of lung volume following any form of lung radiotherapy. With SABR, this "volume reduction" is achieved with a far lower risk of morbidity - in particular, less risk of pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

Pulmonary Function:

* Severe COPD with severe reduction in quality of life due to dyspnea
* Moderate to Severe emphysematous destruction of lung parenchyma on chest CT

  * FEV1 < 45% predicted and >18% predicted
  * FEV1/FVC < .7
  * DLCO > 18% predicted
  * Residual Volume > 160% predicted (by plethysmography)

Arterial Blood Gas:

* paO2>40 on room air at rest
* paCO2<55

General:

* Successful completion of 16 sessions of pulmonary rehabilitation

Exclusion Criteria:

* Predominate chronic bronchitis (none or mild emphysematous destruction of lung on chest CT).
* Pulmonary function tests / lung volumes that do not meet above criteria.
* Active coronary ischemia (stress test required if clinical symptoms).
* Inability to complete 16 sessions of pulmonary rehabilitation.
* Pregnancy.
* Presence of lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Shrager, M.D, Study Director — Stanford University
Locations (1):
- Stanford Cancer Center, Palo Alto, California, United States

REFERENCES:
- [Result] Kamtam DN, Binkley MS, Kapula N, Sadeghi C, Nesbit S, Guo HH, Chang J, Maxim PG, Diehn M, Loo BW Jr, Shrager JB. First in Human Phase 1 Clinical Trial of Stereotactic Irradiation to Achieve Lung Volume Reduction (SILVR) in Severe Emphysema. Int J Radiat Oncol Biol Phys. 2024 Oct 1;120(2):345-356. doi: 10.1016/j.ijrobp.2024.03.049. Epub 2024 Apr 12. PMID 38615887

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants signed consent; 8 were allocated to the study arm.
Groups:
- Stereotactic Ablative Radiotherapy: Stereotactic Ablative Radiotherapy (SABR): 45 Gy in three fractions of 15 Gy, on each side that is treated.
Period: Overall Study
Arm/Group | Stereotactic Ablative Radiotherapy
Started | 9
Received SABR Treatment | 8
Completed | 4
Not Completed | 5
Not completed — Death prior to intervention | 1
Not completed — Death following intervention | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants who received SABR
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 73.0 [63.0 to 78.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients With Grade 3 or Higher Adverse Events.
Description: Adverse events will be based upon National Cancer Institute Common Terminology Criteria
Time Frame: 18 months
Population: Participants who received SABR
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
Participants | 3

2. Secondary Outcome: Change From Baseline Value in Forced Expiratory Volume Percent Predicted
Description: Forced Expiratory Volume will be taken both prior (baseline) and following the procedure (months 6, 12, and 18)
Time Frame: Baseline and months 6, 12, and 18
Population: Participants who received SABR and with data at each respective time point
Measure: Median (Full Range); unit: percentage of predicted value
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
percentage of predicted value
  Baseline | 28.5 [19.0 to 42.0]
  Change at 6 months | 5.0 [-3.0 to 18.0]
  Change at 12 months: number analyzed (Participants) | 3
  Change at 12 months | 3.0 [3.0 to 10.0]
  Change at 18 months: number analyzed (Participants) | 4
  Change at 18 months | 5.5 [-2.0 to 6.0]

3. Secondary Outcome: Change From Baseline Value in Forced Expiratory Volume in 1 Second (Liters)
Description: Forced Expiratory Volume will be taken both prior (baseline) and following the procedure (months 6, 12, and 18)
Time Frame: Baseline and months 6, 12, and 18
Population: Participants who received SABR and with data at each respective time point
Measure: Median (Full Range); unit: liters
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
liters
  Baseline | 0.79 [0.53 to 1.29]
  Change at 6 months | 0.13 [-0.08 to 0.50]
  Change at 12 months: number analyzed (Participants) | 3
  Change at 12 months | 0.14 [-0.03 to 0.25]
  Change at 18 months: number analyzed (Participants) | 4
  Change at 18 months | 0.02 [-0.06 to 0.15]

4. Secondary Outcome: Change From Baseline in Diffusing Capacity for Carbon Dioxide (% Predicted)
Description: Diffusing Capacity for Carbon Dioxide will be taken both prior (baseline) and following the procedure (months 6, 12, and 18)
Time Frame: Baseline and months 6, 12, and 18
Population: Participants who received SABR and with data at each respective time point
Measure: Median (Full Range); unit: percentage of predicted value
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
percentage of predicted value
  Baseline | 40.0 [24.0 to 67.0]
  Change at 6 months | -8.0 [-20.0 to 11.0]
  Change at 12 months: number analyzed (Participants) | 3
  Change at 12 months | -10.0 [-14.0 to 9.0]
  Change at 18 months: number analyzed (Participants) | 4
  Change at 18 months | -3.5 [-22.0 to 11.0]

5. Secondary Outcome: Change From Baseline in 6 Minute Walk Test (Meters)
Description: The walk test will be done both prior (baseline) and following the procedure (month 6)
Time Frame: Baseline and month 6
Population: Participants with available data
Measure: Median (Full Range); unit: meters
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 6
meters
  Baseline | 289.0 [48.0 to 430.0]
  6 months | 406.0 [79.0 to 629.0]
  Change at 6 months | 27.0 [11.0 to 301.0]

6. Secondary Outcome: Total Lung Capacity (% of Predicted Value)
Description: Total Lung Capacity will be measured both prior (baseline) and following the procedure (up to 18 months)
Time Frame: Baseline and date of last available time-point in follow-up period (up to 18 months)
Population: Participants who received SABR and with data at last available time-point in follow-up period
Measure: Median (Full Range); unit: percentage of predicted value
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 6
percentage of predicted value
  Baseline | 127.5 [117 to 146]
  Last available time-point in follow-up period: number analyzed (Participants) | 4
  Last available time-point in follow-up period | 119.5 [104 to 147]

7. Secondary Outcome: Residual Volume (RV) (% of Predicted Value)
Description: Residual volume (RV) is the volume of air remaining in the lungs after maximum forceful expiration. In other words, it is the volume of air that cannot be expelled from the lungs, thus causing the alveoli to remain open at all times.
Time Frame: Baseline and date of last available time-point in follow-up period (up to 18 months)
Population: Participants who received SABR and with data at last available time-point in follow-up period
Measure: Median (Full Range); unit: percentage of predicted value
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
percentage of predicted value
  Baseline | 191 [104 to 255]
  Last available time-point in follow-up period: number analyzed (Participants) | 5
  Last available time-point in follow-up period | 188 [104 to 238]

8. Secondary Outcome: Short Form (SF)-36 Quality of Life Survey Score
Description: The SF-36 Physical Component Summary (PCS) assesses limitations in physical functioning due to health problems, limitations in usual role because of physical health problems, bodily pain, and general health perceptions; the mental component summary (MCS) assesses vitality, limitations in social functioning because of physical or emotional problems, limitations in usual role due to emotional problems, and general mental health. The PCS and MCS scores each range from 0 (worst) to 100 (best). Increases from baseline indicate improvement.
Time Frame: Baseline and months 6
Population: Participants who received SABR and with data at each respective time point
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 8
score on a scale
  PCS-Baseline | 31.9 [24.1 to 43.8]
  PCS-6 months: number analyzed (Participants) | 7
  PCS-6 months | 24.9 [21.1 to 48.6]
  MCS-baseline | 48.0 [21.0 to 58.3]
  MCS-6 months: number analyzed (Participants) | 7
  MCS-6 months | 51.5 [34.6 to 57.9]

9. Secondary Outcome: Modified Borg Dyspnea Scale
Description: This is a patient-reported scale to rate the difficulty of breathing. The scale ranges from 0 to 10, wherein "0" indicates no difficulty breathing, and "10" indicates a maximal difficulty in breathing. Patients may report in whole numbers, from 0 to 10, in addition to reporting 0.5, which indicates "very, very slight (just noticeable) difficulty in breathing."
  A negative change in score indicates a reduction in patient-reported breathing difficulty. The greater the negative change, the better the patient-reported breathing.
Time Frame: Baseline and months 6, 12, and 18
Population: Data were not collected for this outcome measure
Arm/Group | Stereotactic Ablative Radiotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Stereotactic Ablative Radiotherapy
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Ablative Radiotherapy (N=9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 — Possibly related to treatment
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Possibly related to treatment
Heart failure (Cardiac disorders) | 1 — Possibly related to treatment
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Unrelated to treatment
Heart failure (Cardiac disorders) | 1 — Unrelated to treatment
Atrial fibrillation (Cardiac disorders) | 1 — Unrelated to treatment
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — Unrelated to treatment
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 — Unrelated to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Ablative Radiotherapy (N=9)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 — Related to treatment
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 — Unrelated to treatment
Atrial fibrillation (Cardiac disorders) | 1 — Unrelated to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT03673176/Prot_000.pdf